CLINICAL TRIAL: NCT07402343
Title: A Single Arm Phase II Study Evaluating Intracranial Efficacy of Tarlatamab in Patients With Asymptomatic Active Brain Metastases From Small Cell Lung Cancer
Brief Title: Tarlatamab for SCLC Brain Metastases
Acronym: T-BRAIN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other); Erasmus Medical Center (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-BRAIN; 2025-522162-75-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-15; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer; Brain Metastases, Adult
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tarlatamab (Experimental): Tarlatamab intravenous: 1 mg on day 1, followed by 10 mg on days 8 and 15 of cycle 1; thereafter every 2 weeks in cycles of 28 days
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Cycle 1: 1 mg on day 1, followed by 10 mg on days 8 and 15 Cycles thereafter: 10 mg every two weeks, in cycles of 28 days Treatment continues till unacceptable toxicity or disease progression

SUMMARY:
A single arm phase II study evaluating intracranial efficacy of tarlatamab in patients with asymptomatic active brain metastases from small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
Patients with small cell lung cancer (SCLC) have a high risk of brain metastases (BM). Due to the decline in the use of prophylactic cranial irradiation (PCI), because of the risk of toxicity in absence of a survival benefit, as well as increased imaging follow-up, the incidence of BM in SCLC will rise compared to the PCI-era. Upon central nervous system (CNS) progression on first line therapy, cranial radiotherapy can be given but effect is modest. All standard of care second line drugs have limited (prolonged) efficacy in the CNS, or efficacy is unknown. Therefore, new systemic therapies that are active systemically as well as intracranially are needed.

Tarlatamab is a bispecific T-cell engager targeting delta-like ligand 3 (DLL3) and CD3 and has shown promising activity in heavily pretreated patients with SCLC. With a median follow-up of 20.7 months, objective response rate (ORR) was 40% in a phase II trial, DCR was 70%, median PFS was 4.3 months, median OS 15.2 months and 26% had sustained disease control ≥52 weeks. The most common adverse event was cytokine release syndrome (CRS, 53% in the 10 mg group), with the majority being grade 1-2, and 1% grade 3. Similar long-term follow-up data was reported for the phase I trial. CNS disease progression occurred in only 9/112 enrolled patients (25% had baseline BM).

Seventeen patients with previously treated BM with a size of ≥ 10mm were enrolled. Modified Response Assessment in Neuro-Oncology (RANO) criteria showed CNS tumor shrinkage ≥30% in 59% (10/17) of these patients, and intracranial disease control in 94%. Out of the 10 patients with CNS tumor shrinkage of ≥30%, five had cranial radiotherapy >5 weeks before the start of tarlatamab, which indirectly indicates that tarlatamab could have intracranial activity. Additionally, the confirmatory randomized phase III trial DeLLphi-304 (NCT05740566) enrolling patients with relapsed SCLC and randomizing between tarlatamab and standard of care chemotherapy was positive for its primary outcome, OS. Median OS was 13.6 months for tarlatamab and 8.3 months for standard of care (hazard ratio 0.60, 95% confidence interval 0.47-0.77, p <0.001). Additionally, tarlatamab resulted in a PFS benefit as well as less treatment related toxicity. Moreover, patients with (treated) BM derived at least the same magnitude of benefit (HR for OS with baseline BM 0.45, HR for OS if no baseline BM 0.81). At the end of the enrollment, the protocol was amended to allow patients with asymptomatic untreated BM. However, meaningful data regarding CNS efficacy of tarlatamab will not be obtained in this study. Therefore, it is of interest to evaluate tarlatamab in patients with SCLC with disease progression including BM on first line systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Signed and written informed consent
2. Age 18 years or older
3. Patients with pathology proven metastatic SCLC
4. Pretreated with at least platinum-doublet chemotherapy with or without immunotherapy, no maximum of previous lines of systemic therapy
5. WHO/ECOG PS 0-1
6. Estimated life expectancy 12 weeks or more
7. At least one asymptomatic active (newly diagnosed or unequivocally progressive) untreated brain metastasis ≥ 5mm:

   1. Subjects with largest measurable intracranial lesion ≥5 mm but <10mm may be allowed to enroll upon agreement with investigator (for patients with target lesions of ≥ 5mm but <10 mm, 1.5 mm slice thickness brain MRI is required).
   2. "Untreated" refers to the lesion not being previously treated with stereotactic radiosurgery/therapy (SRS/SRT) or surgery.
   3. Prior treatment with whole brain radiation therapy or local surgery is permissible provided unequivocal progression in the lesion has since occurred
8. For at least 7 days prior to study start: Patient must be asymptomatic from CNS metastases and on a stable dose of anti-epileptics and corticosteroids. Maximum dose of steroids is 10 mg prednisolone or equivalent/day, dose should be noted.
9. Adequate organ and bone marrow function, defined as:

   a. Hematological function: i. Absolute neutrophil count ≥1.5 x109/L ii. Platelet count ≥ 100 x109/L iii. Hemoglobin ≥ 5.6 mmol/l b. Coagulation function: i. Protrombin time (PT)/ international normalized ratio (INR) and partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) ≤ 1.5 x institutional upper limit of normal (ULN) except for subjects receiving anticoagulation, who must be on a stable dose of anticoagulant therapy for 6 weeks prior to start of study treatment.

   c. Renal function: i. Estimated glomerular filtration rate (eGFR) based on Modification of Dietin Renal Disease (MDRD) calculation > 30 mL/min/1.73 m2 d. Hepatic function: i. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3x ULN (or < 5x ULN for subjects with liver metastases) ii. Total bilirubin < 1.5x ULN (or < 2x ULN for subjects with liver metastases), except for subjects with Gilberts disease e. Pulmonary function: i. No clinically significant pleural effusion. Pleural effusions managed with indwelling pleural catheter (eg, PleurX) are allowed.

ii. Baseline oxygen saturation > 90% on room air f. Cardiac function: i. Cardiac ejection fraction ≥50%, no clinically significant pericardial effusion as determined by an echocardiogram (ECHO) or multigated acquisition (MUGA) scan, and no clinically significant electrocardiogram (ECG) finding

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Symptomatic BM (if asymptomatic with corticosteroids with a maximum dose of steroids of 10 mg prednisolone or equivalent/day, the patient is eligible). If in doubt, discussion with the sponsor is necessary
2. Leptomeningeal metastases (evaluated with MRI brain)
3. BM in eloquent area (to be discussed with neuro-oncologist)
4. Contra-indication for MRI
5. Prior history of severe or life-threatening events from any immune-mediated therapy
6. Grade 2 or higher toxicity from previous systemic therapy, except for alopecia
7. History of other malignancy within the past 2 years, with the following exceptions:

   1. Malignancy treated with curative intent before enrolment, with no known active disease and felt to be at low risk for recurrence by the treating physician, after discussion with the sponsor
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. adequately treated cervical cancer in situ without evidence of disease
   4. adequately treated breast ductal carcinoma in situ without evidence of disease
   5. prostatic intraepithelial neoplasia without evidence of prostate cancer
   6. adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], systemic lupus erythematosus, sarcoidosis, granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc), autoimmune pneumonitis, and autoimmune myocarditis. The following are exceptions to this criterion:

   1. Subjects with vitiligo or alopecia
   2. Subjects with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Subjects without active disease in the last 5 years may be included but only after consultation with the sponsor
   5. Subjects with coeliac disease controlled by diet alone
9. Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II, appendix 2), within 6 months prior to first dose of study treatment
10. History of arterial thrombosis (e.g. stroke or transient ischemic attack) within 6 months prior to first dose of study treatment
11. Evidence of ILD or active, non-infectious pneumonitis
12. History of solid organ transplant
13. Major surgical procedures within 28 days prior to first dose of study treatment
14. Presence of active HIV or hepatitis infection

    1. HIV infection: subjects with HIV infection on antiviral therapy and undetectable viral load are permitted with a requirement for regular monitoring for reactivation for the duration of the treatment on study per local or institutional guidelines
    2. Active hepatitis C infection (subjects with detectable hepatitis C antibody [HCV Ab] and hepatitis C virus (HCV) RNA viral load above the limit of quantification) are not allowed. Subjects with presence of HCV antibody (HCV Ab positive) and HCV RNA viral load below the limit of quantification (HCV RNA negative) with or without prior treatment are allowed
    3. Active hepatitis B infection (subjects with presence of hepatitis B surface antigen [HBsAg-positive] and hepatitis B virus (HBV) DNA viral load above the limit of quantification [HBV DNA positive) are not allowed. Subjects with resolved HBV infection, defined as absence of HBV surface antigen (HBsAg-negative) and presence of HBV core antibody (anti-HBc positive) followed by an HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines. Subjects with inactive HBV infection inactive carrier state, defined as presence of HBV surface antigen (HBsAg-positive) and HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed with the requirement for regular monitoring for reactivation for the duration of the treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
15. Receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 14 days prior to first dose of study treatment

    a. Low-dose corticosteroids (prednisone ≤ 10 mg per day or equivalent is permitted during the study)
16. Subjects with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment

    a. Note: simple urinary tract infection and uncomplicated bacterial pharyngitis are permitted if responding to active treatment. Subjects requiring oral antibiotics who have been afebrile > 24 hours, have no leukocytosis, nor clinical signs of an infection are eligible. Screening for chronic infectious conditions is not required unless otherwise noted as exclusion criteria.
17. Treatment with live virus, including live-attenuated vaccination, within 4 weeks prior to the first dose of study treatment. Inactive vaccines (e.g. non-live or non-replication agent) and live viral non-replicating vaccines (e.g. Jynneos for mpox infection) within 3 days prior to first dose of study treatment
18. Prior therapy with any selective inhibitor of the DLL3 pathway
19. Receiving another anticancer therapy. Adjuvant hormonal therapy for resected breast cancer is permitted.
20. Treatment in an alternative investigational trial within 28 days prior to enrollment
21. Female subjects of childbearing potential unwilling to use protocol specified method of contraception (appendix 3) during treatment and for an additional 60 days after the last dose of tarlatamab
22. Female subjects who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of tarlatamab
23. Female subjects planning to become pregnant or donate eggs while on study through 60 days after the last dose of tarlatamab
24. Female subjects of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive serum pregnancy test
25. Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 60 days after the last dose of tarlatamab
26. Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of tarlatamab
27. Male subjects unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of tarlatamab
28. Subject has known sensitivity to any of the products or components to be administered during dosing of tarlatamab.
29. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
30. Subjects likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigators knowledge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Intracranial overall response rate (ORR) | Up to 36 months
  Brain metastases ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on central and local investigator's assessment according to RANO-BM criteria on brain MRI

SECONDARY OUTCOMES:
Brain metastases (BM) disease control rate (DCR) and median CNS PFS | Up to 36 months
  DCR is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Non-CR/Non-PD according to RANO-BM on brain MRI
Extracranial ORR and DCR | Up to 36 months
  Extracranial ORR and DCR is evaluated according to RECIST 1.1, measured with CT.
  ORR is defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment, DCR is defined as the proportion of participants with Best Overall Response (BOR) of CR, PR, Stable Disease (SD) or Non-CR/Non-PD.
Extracranial PFS | Up to 36 months
  Extracranial progression free survival (PFS) will be assessed according to RECIST 1.1 based on CT.
  PFS is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause.
Overall PFS | Up to 36 months
  Overall progression free survival (PFS) is evaluated according to RECIST 1.1 based on CT for extracranial lesions, and RANO-BM based on MRI for BM.
Overall survival | Up to 48 months
  Overall survival (OS) is defined as the time from date of start of treatment to date of death due to any cause
Number of patients experiencing adverse events according to CTCAE and ASTCT criteria | Up to 36 months
  Number of patients experiencing adverse events, according to ASTCT 2019 criteria for immuno effector cell-associated neurotoxicity syndrome (ICANS) and cytokine release syndrome (CRS), and according to CTCAE v5.0 for other adverse events.

OTHER OUTCOMES:
Efficacy of tarlatamab in relation to previous cranial radiotherapy | Up to 36 months
  Exploratory endpoint: comparison of the efficacy of tarlatamab in patients who previously received cranial radiotherapy to the efficacy in those who were not previously treated with cranial radiotherapy
Safety of tarlatamab in relation to previous cranial radiotherapy | Up to 36 months
  Exploratory endpoint: comparison of the safety of tarlatamab in patients who previously received cranial radiotherapy to the safety of tarlatamab in those who were not previously treated with cranial radiotherapy
Efficacy of tarlatamab in relation to concomitant steroid use | Up to 36 months
  Exploratory endpoint: comparison of the efficacy of tarlatamab in patients who concomitantly used steroids to the efficacy in those who were not concomitant steroid users.
Safety of tarlatamab in relation to concomitant steroid use | Up to 36 months
  Exploratory endpoint: comparison of the safety of tarlatamab in patients who concomitantly used steroids to the safety in those who were not concomitant steroid users.
Evaluate immune environment in cerebrospinal fluid (with lumbar puncture) versus peripheral blood in relation to SCLC responses | Up to 36 months
  Exploratory endpoint:
  tumor response (BM and extracranial response, such as progressive disease, stable disease or (partial) response) in relation to baseline and 12 week evaluation of immune cells in liquor and peripheral blood, respectively.
  Lumbar puncture not mandatory

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - The Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen
  - Maastricht UMC+, Maastricht
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No